CLINICAL TRIAL: NCT01995916
Title: Intervention for Menstrual Mood Disorders & Early Life Abuse: BioPsych Mechanisms
Brief Title: Wellness Intervention for Menstrual Mood Disorders
Acronym: WIMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-1867; 1R01MH099076-01A1 (NIH)
Record Dates: First submitted 2013-11-07; First posted 2013-11-27 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Menstrual Mood Disorders
MeSH Terms: interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Intervention (Experimental): Mindfulness Based Stress Reduction Intervention
  Interventions: Behavioral: Mindfulness Intervention
- Social Support Group (Active Comparator): Social Support Group Intervention
  Interventions: Behavioral: Social Support Group

INTERVENTIONS:
Behavioral: Mindfulness Intervention — The Mindfulness Group will meet once a week for 2.5 hours for 8 weeks with a half day retreat.
  Arms: Mindfulness Intervention
Behavioral: Social Support Group — The Social Support Group will meet once a week for 2.5 hours for 8 weeks with a half day retreat.
  Arms: Social Support Group

SUMMARY:
This study has been funded by National Institute of Mental Health (NIMH) to compare two behavioral interventions for Menstrual Mood Disorders, including premenstrual dysphoric disorder (PMDD). Both of these interventions will be run in a group format, meaning that you will be part of a group of other women who have a menstrual mood disorder. Both of these interventions will be run by experienced mental health professionals and both interventions have been shown to be effective in reducing mood symptoms, increasing a sense of well-being, and helping individuals cope with stress. While it is expected that both interventions to be associated with some benefit, this study is designed to see which is better for women with a menstrual mood disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meets prospective criteria for a menstrual mood disorder, including PMDD
* Depression symptom severity and functional impairment based on prospective symptom ratings for 2-3 cycles using the Daily Record of Severity of Problems (DRSP)
* Clear remission of all symptoms during days 6-10
* 18 - 55 years of age
* Regular menstrual cycles
* Early life sexual or physical abuse (50% of sample) or no history of sexual or physical abuse (50% of sample)
* Absence of current PTSD symptoms using the 17-item PTSD checklist (PCL)
* 8th grade literacy level
* Ability to give informed consent

Exclusion Criteria:

* Current Axis I disorder or suicide ideation (histories of depression, anxiety, substance abuse, and eating disorders are allowed if in remission for >2 years)
* Premenstrual exacerbation of chronic disorders
* In a current abusive relationship or residing with a former abuser
* A lifetime history of suicide attempt, or suicidal thoughts or gestures within 5 years of study enrollment
* Histories of bipolar or psychotic disorders
* Age < 18 or > 55 years
* Pregnancy or breastfeeding
* Use of psychotropic, hormonal or other agents that alter mood or biological mediators
* Current functional pain disorder
* A history of meditation practice (2+ times/week for 15+ min; some yoga allowed)
* Diabetes
* BMI < 18.5
* Vigorous exercise
* Stage 2 Hypertension
* Any symptom item rated >2 (moderate or higher) or a total score > 24 on the PTSD checklist

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Premenstrual Depression Symptomatology and Functional Impairment | Baseline, 8 weeks intervention, 6 months follow up
  Premenstrual depression symptoms will be assessed prospectively before, during and for 6 months after the intervention using Daily Record of Severity of Problems (DRSPs). Functional impairment will be assessed via questionnaire at baseline, at 2 week intervals throughout the intervention, and monthly during the follow-up phase.
Change in Cold Pain Sensitivity | Lab 1 before the start of the intervention, Lab 2 immediately following intervention, Labs 3 and 4 during month 3 and 6 of follow up phase
  Sensitivity to a cold pressor pain test (hand submerged in ice water) will be assessed in a laboratory setting before and after the intervention, and again 3 and 6 months later

SECONDARY OUTCOMES:
Change in premenstrual anxiety, irritability and total symptom severity | Baseline, 8 weeks intervention, 6 months follow up
  Symptoms will be assessed prospectively through Daily Record of Severity of Problems (DRSPs).
Change in sensitivity to the temporal summation of heat pain test | Lab 1 before the start of the intervention, Lab 2 immediately following intervention, Labs 3 and 4 during month 3 and 6 of follow up phase
  Sensitivity to a temporal summation of heat pain test will be assessed in a laboratory setting before and after the intervention, and again 3 and 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Susan Girdler, PhD, Principal Investigator — UNC- Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Andersen E, Geiger P, Schiller C, Bluth K, Watkins L, Zhang Y, Xia K, Tauseef H, Leserman J, Girdler S, Gaylord S. Effects of Mindfulness-Based Stress Reduction on Experimental Pain Sensitivity and Cortisol Responses in Women With Early Life Abuse: A Randomized Controlled Trial. Psychosom Med. 2021 Jul-Aug 01;83(6):515-527. doi: 10.1097/PSY.0000000000000889. PMID 33259351